CLINICAL TRIAL: NCT02813278
Title: Efficacy of Simo Decoction and Acupuncture or Chewing Gum Alone on Postoperative Ileus in Colorectal Cancer Resection: a Randomized Clinical Trial
Brief Title: Simo Decoction and Acupuncture on POI in Colorectal Cancer
Acronym: SMD/POI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yang Yang, Le-Qun Li, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMD/POI
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- simo decoction and acupuncture with vitamin B1 (Experimental): Patients will receive simo decoction (10 mL/piece,three times per day) and bilateral tsusanli acupoint injections with vitamin B1 two times per day, starting in the first day after resection for 5 days or until flatus.
  Interventions: Dietary Supplement: simo decoction
- gum chewing (Active Comparator): Patients will receive gum chewing (three times per day) in the first day after resection for 5 days or until flatus.
  Interventions: Other: gum chewing
- empty control (No Intervention): Patients only receive best support care.

INTERVENTIONS:
Dietary Supplement: simo decoction — Participants allocated to SMD and acupuncture were asked to take oral SMD decoction (Hansen Co., Ltd., Yiyang, Hunan province, China, 10 mL/dose) three times per day beginning on the first day after colorectal resection. They also received bilateral injections of vitamin B1 (50 mg x 2) at the tsusanli acupoint one time per day. This intervention was performed for a total of 5 consecutive days or until flatus.
  Arms: simo decoction and acupuncture with vitamin B1
Other: gum chewing — Participants allocated to chewing gum were instructed to chew commercially available sugar-free gum (Extra & Reg, Wm. Wrigley Jr. Co., Ltd., Shanghai, China) three times daily starting on the first postoperative morning. They were instructed to chew the piece of gum for at least 10 min. This intervention was performed for 5 consecutive days or until flatus.
  Arms: gum chewing

SUMMARY:
Colorectal cancer resection is one of the most common types of abdominal surgery. Though most patients undergoing colorectal resection show recovery of bowel movements within a week, some have prolonged intestinal paralysis or postoperative ileus, resulting in decreasing patient comfort, increasing morbidity and mortality, a longer hospital stay and subsequent increased healthcare costs.

DETAILED DESCRIPTION:
Prevention the incidence of postoperative ileus (POI) is quite important because of the negative clinical outcomes it causes. In the past two decades, many treatments and care approaches, such as fluid restriction, early enteral nutrition, and nonsteroidal anti-inflammatory drug are used for the management of POI. In theory of traditional Chinese medicine, oral simo decoction (SMD) or acupuncture at the tsusanli acupoint can boost gastrointestinal hypomotility. The efficacy of accelerating the return of gastrointestinal function by such single method or combination of them has been validated in randomized controlled trials and systematic review following several types of surgery. In recent years, chewing gum, a new and simple modality, has become a commonly applied method in order to prevent and reduce the POI. Systematic reviews and meta-analyses revealed that chewing gum provided significant benefits for the improvement of postoperative bowel function. More importantly, many official guidelines recommend chewing gum for an evidence-based approach in the prevention of POI. Despite these positive evidence, three newest randomized controlled trials are unable to demonstrate an effect of chewing gum on the recovery of bowel function after colorectal resection.

It is important to note that almost all previous randomized controlled trials are based on small sample size. This raises the question whether postoperative SMD, acupuncture at the tsusanli acupoint, or chewing gum can reduce risk of POI following colorectal resection among patients with large sample size. To examine this question, we conducted this randomized controlled trial to compare incidence of POI and length of hospital stay in colorectal cancer patients who received SMD and acupuncture, chewing gum or no intervention following resection.

ELIGIBILITY:
Inclusion Criteria:

* Underwent open or laparoscopic colorectal cancer resection
* Diagnosis of colorectal cancer was confirmed by histopathological examination of surgical samples in all patients

Exclusion Criteria:

* Previously underwent exploratory laparotomy
* Known Central Nervous System tumors including metastatic brain disease
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
First flatus time | one day
Length of hospital stay | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Yang Yang, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Heijkant TC, Costes LM, van der Lee DG, Aerts B, Osinga-de Jong M, Rutten HR, Hulsewe KW, de Jonge WJ, Buurman WA, Luyer MD. Randomized clinical trial of the effect of gum chewing on postoperative ileus and inflammation in colorectal surgery. Br J Surg. 2015 Feb;102(3):202-11. doi: 10.1002/bjs.9691. Epub 2014 Dec 18. PMID 25524125
- [Background] Kobayashi T, Masaki T, Kogawa K, Matsuoka H, Sugiyama M. Efficacy of Gum Chewing on Bowel Movement After Open Colectomy for Left-Sided Colorectal Cancer: A Randomized Clinical Trial. Dis Colon Rectum. 2015 Nov;58(11):1058-63. doi: 10.1097/DCR.0000000000000452. PMID 26445178
- [Background] Atkinson C, Penfold CM, Ness AR, Longman RJ, Thomas SJ, Hollingworth W, Kandiyali R, Leary SD, Lewis SJ. Randomized clinical trial of postoperative chewing gum versus standard care after colorectal resection. Br J Surg. 2016 Jul;103(8):962-70. doi: 10.1002/bjs.10194. Epub 2016 May 5. PMID 27146793
- [Derived] Yang Y, Zuo HQ, Li Z, Qin YZ, Mo XW, Huang MW, Lai H, Wu LC, Chen JS. Comparison of efficacy of simo decoction and acupuncture or chewing gum alone on postoperative ileus in colorectal cancer resection: a randomized trial. Sci Rep. 2017 Jan 19;7:37826. doi: 10.1038/srep37826. PMID 28102199